CLINICAL TRIAL: NCT06269705
Title: A Study to Evaluate the Efficacy and Safety of ZILRETTA in Subjects With Glenohumeral Osteoarthritis
Brief Title: ZILRETTA in Subjects With Shoulder Osteoarthritis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 006-C-301
Record Dates: First submitted 2024-02-13; First posted 2024-02-21 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Glenohumeral Osteoarthritis
Keywords: Glenohumeral Osteoarthritis
MeSH Terms: interventions — Triamcinolone; Saline Solution

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Only unblinded team (pharmacist, unblinded coordinator, drug administrator) will know the treatment assignment. A site-specific blinding plan will be developed to ensure blinding. Unblinded team will only interact with the subject at treatment and will not have any blinded roles on the study (only exception- informed consent). The subject and the assessor responsible for assessments/safety monitoring will be blinded. Site and Sponsor personnel/representatives will be blinded, with the following Sponsor/representative exceptions: unblinded monitors for performing drug accountability, unblinded clinical manager for reviewing unblinded monitoring visit reports and escalation of site unblinded issues, inventory manager for addressing product-related issues, and regulatory personnel for safety reporting. Information regarding treatment assignments will be kept securely at Sponsor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ZILRETTA (Experimental): 100 subjects will receive 32 mg ZILRETTA
  Interventions: Drug: ZILRETTA
- Placebo (Placebo Comparator): 50 subjects will receive normal saline placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: ZILRETTA — IA injection of 32 mg ZILRETTA
  Arms: ZILRETTA
Other: Placebo — IA injection of placebo (normal saline)
  Other Names: Normal Saline
  Arms: Placebo

SUMMARY:
Primary Objective: To assess the efficacy of ZILRETTA on pain following an intra-articular (IA) injection in subjects with glenohumeral osteoarthritis (OA) relative to normal saline placebo

Secondary Objective:

* To assess the efficacy of ZILRETTA on pain following an IA injection in subjects with glenohumeral OA relative to triamcinolone acetonide injectable suspension, and normal saline placebo
* To assess the safety of ZILRETTA in subjects with glenohumeral OA relative to normal saline placebo

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind, parallel-group study to evaluate the efficacy and safety of ZILRETTA in subjects with glenohumeral OA. This study will be conducted at approximately 25 study sites in the United States. Subjects will be screened to confirm the diagnosis of OA and eligibility based on the Inclusion and Exclusion Criteria. Approximately 150 male or female subjects, 50 to 80 years of age inclusive, will be enrolled, randomized to 1 of 2 treatment groups (2:1), and treated with a single IA injection of either:

* Treatment Arm: 32 mg ZILRETTA,
* Treatment Arm: placebo (normal saline). ZILRETTA, or normal saline placebo will be administered as a single IA injection with a 24-week follow-up period with a primary endpoint at Week 12.

The study will involve a Screening period (a minimum of 10 days, up to a maximum of 35 days), pre-treatment phase, dosing at Baseline/Day 1, and 8 additional outpatient visits at Weeks 2, 4, 8, 12, 16, 20, and 24/End of Study (EOS) during the study.

At specified times throughout the study, subjects will undergo physical examinations, index shoulder assessments, and index shoulder X-rays; blood will be collected for laboratory safety tests; and vital signs will be collected.

Information regarding adverse events (AEs) and prior and concomitant medications and treatments will be collected from the time of signing the Informed Consent Form (ICF) through the Week 24/EOS visit. Information regarding rescue medication usage, Average and Worst daily Pain score (0-10 Numeric Rating Scale (NRS); 0 = no pain, 10 = worst possible pain) in the index shoulder, and Sleep Interference (SI) will be completed daily via an electronic diary (eDiary) and reviewed for compliance by site staff at each study visit.

At the Screening Visit, subjects will be registered in the eDiary and receive instructions on its use. Subjects will complete accurate pain reporting (APR) and placebo response reduction (PRR) training prior to completing all questionnaires.

ELIGIBILITY:
Inclusion Criteria

To be included in the trial, participants must fulfill the following criteria:

1. Written informed consent has been obtained prior to initiating any study-specific procedures.
2. Willingness and ability to comply with the study procedures and visit schedules and ability to follow verbal and written instructions, including eDiary questionnaire completion requirements.
3. Participants 50 to 80 years of age, inclusive, on the day of consent.
4. Body mass index (BMI) does not prohibit proper identification of bony landmarks and/or otherwise prohibit the ability to properly inject into the shoulder joint per Principal Investigator's (PI's) judgment.
5. Participants with shoulder pain and glenohumeral arthritis with or without rotator cuff pathology (eg, rotator cuff inflammation, partial rotator cuff tear [non-to-mild superior subluxation of the humeral head on X-ray] may be included). Participants with positive Neer and Hawkins-Kennedy tests on index shoulder exam should be excluded. Participants who have complete or irreparable rotator cuff tear should not be included.
6. Grade 1, 2, or 3 OA in the index glenohumeral joint based on the Samilson-Prieto classification system as confirmed by X-ray (axillary view and true anterior-posterior view) taken at, or within 6 months of, the Screening Visit and read by the central reader.
7. Average daily mean pain score ≥4.0 and ≤9.0 in index shoulder (0-10 numeric rating scale [NRS]) using the average daily ratings for at least 4 out of the 7 days prior to Baseline/Day 1.
8. Average Shoulder Pain and Disability Index (SPADI) pain score ≥4.0 and ≤9.0 in index shoulder during the Screening and Pretreatment Phase (average score) as calculated and reported in the electronic Clinical Outcomes Assessment (eCOA).
9. Willingness to abstain from use of protocol-specified restricted medications and therapies during the study.
10. Sexually active males or females of childbearing potential must agree to use a highly effective method of contraception throughout the duration of the study. Females of childbearing potential are defined as females who are not surgically sterile or postmenopausal (defined as 12 consecutive months with no menses without an alternative medical cause) as documented in medical history. Highly effective methods of contraception include abstinence; oral, injected, or implanted hormonal methods of contraception; intrauterine device or intrauterine system; condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository; or monogamous intercourse with a partner who is surgically sterile (post-vasectomy, -hysterectomy, or -tubal ligation).

Exclusion Criteria

Participants fulfilling at least 1 of the following criteria may not be included in the study:

Disease-Related Criteria

1. Participants who cannot washout prohibited medications (eg, opioids, other analgesics, and tetrahydrocannabinol (THC)- and cannabidiol (CBD)-containing products) or restricted medications.
2. Has symptomatic arthritis in other joints of the index shoulder (eg, acromioclavicular joint, sternoclavicular joint, or pain in the scapulothoracic region), which is the primary source of pain in the opinion of the Investigator.
3. Has clinical symptomatic chronic bilateral shoulder pain (any condition causing pain in the non-index shoulder).
4. Has a subchondral bone insufficiency fracture or humeral head necrosis/collapse (including bone infarct) in the index shoulder based on X-ray used for study qualification.
5. Has a prior ipsilateral proximal humerus fracture or scapula fracture to the index shoulder within 2 years of Screening Visit.
6. Has current diagnosis of adhesive capsulitis ("frozen shoulder") in the index shoulder or previous diagnosis within 1 year of the Screening Visit and is still not resolved.
7. Has a previous substantial shoulder injury or trauma (eg, glenohumeral dislocation or clavicle fracture) in the index shoulder which resulted in functional limitation within 3 months prior to the Screening Visit.
8. Has had prior surgery on the index shoulder (less than 3 years), either open or arthroscopic. Should not have any retained hardware.
9. Has an index shoulder with major dysplasia or congenital abnormality, osteochondritis dissecans, acromegaly, ochronosis, hemochromatosis, Wilson's disease, primary osteochondromatosis, chondrolysis from a pain pump, or a history of avascular necrosis with secondary OA or any other anatomic variation or disease that, in the opinion of the Investigator, could interfere with either the injection procedure or the study outcome.
10. Has current or history of infection (eg, osteomyelitis) in the index shoulder or current skin infection at injection site.
11. Has any concurrent chronic joint, muscle, or nerve pain condition within 1 month prior to the Screening Visit (participant self-report acceptable), including but not limited to, cervical spine pain or conditions causing radicular pain or peripheral nerve injury/entrapment (eg, brachial plexus injury or suprascapular nerve entrapment); diabetic neuropathy of upper extremities; post-herpetic neuralgia; post-stroke pain; or fibromyalgia that may affect sensation of the index shoulder.
12. painDETECT Questionnaire (PD-Q) score >18 during Screening Visit.
13. History or current evidence of reactive arthritis, rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, or arthritis associated with inflammatory bowel disease, systemic lupus erythematosus, or calcium pyrophosphate dihydrate crystal deposition (CPPD), gout, or other autoimmune diseases.
14. Any planned surgeries in the upper limbs and/or cervical spine during the study period, or any other surgery during the study period that would require use of a restricted medication.

    Previous or Concomitant Treatment-Related Criteria
15. Presence of surgical hardware or other foreign body due to open or arthroscopic cartilage transplant or bone grafting procedures in the index shoulder.
16. Use of muscle relaxants (eg, cyclobenzaprine, tetrazepam, and diazepam) or oral/topical therapies (eg, nonsteroidal anti-inflammatory drugs [NSAIDs], CBD oil, capsaicin, lidocaine patches, or other local treatments) applied to the index shoulder within 1 month prior to Screening Visit or within 5 half-lives of last dose.
17. The use of corticosteroids (any route of administration: IA, intrabursal, intratendinous, intravenous [IV], intramuscular [IM], oral, or inhaled) within 3 months of Screening Visit except occasional (non-daily use <1 month) topical and intranasal steroid use within 1 month prior to dosing. Treatment in another joint during this timeframe is exclusionary.
18. IA treatment of index shoulder with any of the following agents within 6 months or 5 half-lives of Screening: hyaluronic acid (investigational or marketed) or any biologic agent (eg, platelet rich plasma [PRP] injection, stem cells, prolotherapy, and amniotic fluid-derived product).
19. Significant changes with regard to physical activity, physical therapy, or lifestyle within 1 month of the Screening Visit, or any planned changes throughout the duration of the study.
20. Use of selective serotonin reuptake inhibitors (SSRIs)/serotonin and norepinephrine reuptake inhibitors (SNRIs) (eg, fluoxetine, fluvoxamine, citalopram, escitalopram, sertraline, duloxetine, and venlafaxine, milnacipran) if the dose is not stable for at least 3 months prior to Screening Visit and must remain stable throughout the study.
21. Any treatment with acupuncture and/or transcutaneous electrical nerve stimulation (TENS) within 3 months of Screening Visit.

    Participant-Related Criteria
22. Females who are pregnant or nursing or plan to become pregnant within 12 months after dosing; men whose partner plans to conceive within 12 months after dosing.
23. Participants with clinically relevant level of pain catastrophizing defined as Pain Catastrophizing Scale (PCS) score of ≥30 at Screening Visit.
24. Known or suspected hypersensitivity to any form of triamcinolone or PLGA.
25. Laboratory evidence of infection with human immunodeficiency virus (HIV), positive test for hepatitis B surface antigen (HBsAg), or positive for hepatitis C virus (HCV) antibodies.
26. A medical history suggesting the participant will or is likely to require a course of systemic corticosteroids during the study.
27. History or evidence of active or latent systemic fungal or mycobacterial infection (including tuberculosis) or of ocular herpes simplex.
28. History of sarcoidosis, amyloidosis, or active Cushing's syndrome.
29. Use of immunomodulators, immunosuppressives, or chemotherapeutic agents within 5 years of Screening.
30. Active or history of malignancy within 5 years of Screening, with the exception of resected basal cell carcinoma, squamous cell carcinoma of the skin, or effectively managed cervical carcinoma.
31. History of radiation treatment involving the index shoulder girdle.
32. Active substance use/abuse (drugs or alcohol) or history of substance abuse within 12 months of Screening. Positive drug test results due to prescribed attention deficit/hyperactivity disorder (ADHD) medications with at least 6 months of stable dosing is permitted.
33. Has received a live vaccine (eg, measles, mumps, and rubella [MMR], rotavirus, yellow fever, varicella, influenza (nasal spray version only), Bacillus Calmette-Guérin [BCG], and polio) within 3 months of Baseline/Day 1.
34. Has received an inactivated vaccination (eg, flu, COVID, tetanus, tetanus/diphtheria/pertussis [Tdap], hepatitis A) within 1 week prior to the Screening Visit and local injection pain has not resolved.
35. Use of any other investigational drug, biologic, or device within 3 months of Screening Visit.
36. Any bacterial or viral infection requiring IV antibiotics within 4 weeks of Baseline/Day 1 or oral antibiotics within 2 weeks of Baseline/Day 1.
37. Any other clinically significant acute or chronic medical conditions (eg, asthma or chronic obstructive pulmonary disease [COPD] requiring steroid use, poorly controlled diabetes with hemoglobin A1c [HbA1c] of greater than 9.5%) that, in the judgment of the Investigator, could compromise participant safety, preclude the use of an IA corticosteroid, limit the participant's ability to complete the study, or compromise the objectives of the study.
38. Participants contraindicated to the use of acetaminophen/paracetamol (allowed rescue pain medicine) per National Product Labeling and Investigator's judgment.
39. Participant is the Investigator or any Subinvestigator, research assistant, pharmacist, study coordinator, or other staff or relative thereof directly involved in the conduct of the study.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline on the Worst Daily Pain (24-hr) mean score (0-10 Numeric Rating Scale (NRS); 0 = no pain, 10 = worst possible pain) at Week 12 for ZILRETTA relative to placebo | Week 12

SECONDARY OUTCOMES:
Change from Baseline on the Worst Daily Pain (24-hr) mean score (0-10 Numeric Rating Scale (NRS); 0 = no pain, 10 = worst possible pain) at Week 12 for ZILRETTA relative to TCA-IR | Week 12
Change from Baseline on the Worst Daily Pain (24-hr) mean score (0-10 Numeric Rating Scale (NRS); 0 = no pain, 10 = worst possible pain) at Week 18 for ZILRETTA relative to TCA-IR | Week 18
Change from Baseline on the Worst Daily Pain (24-hr) mean score (0-10 Numeric Rating Scale (NRS); 0 = no pain, 10 = worst possible pain) at Week 2 for ZILRETTA relative to placebo | Week 2
Change from Baseline on the Worst Daily Pain (24-hr) mean score (0-10 Numeric Rating Scale (NRS); 0 = no pain, 10 = worst possible pain) at Week 4 for ZILRETTA relative to placebo | Week 4
Change from Baseline on the Worst Daily Pain (24-hr) mean score (0-10 Numeric Rating Scale (NRS); 0 = no pain, 10 = worst possible pain) at Week 8 for ZILRETTA relative to placebo | Week 8
Change from Baseline at Week 12 on the Shoulder Pain and Disability Index (SPADI) total score and subscales (0-10 Numeric Rating Scale (NRS); 0 = no pain, 10 = worst possible pain) for ZILRETTA relative to placebo | Week 12
Change from Baseline at Week 12 on the SPADI total score and subscales (0-10 Numeric Rating Scale (NRS); 0 = no pain, 10 = worst possible pain) for ZILRETTA relative to TCA-IR | Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Nino Joy, MD, Study Director — Pacira Pharmaceuticals, Inc
Locations (32):
- United States (32):
  - Alabama Orthopaedic Center- Research, Vestavia Hills, Alabama
  - Onyx Clinical Research, Surprise, Arizona
  - Tucson Orthopaedic Institute (TOI) - East Office, Tucson, Arizona
  - Horizon Clinical Research, La Mesa, California
  - Napa Pain Institute, Napa, California
  - Stanford University - Sports Medicine Clinic, Redwood City, California
  - International Spine, Pain & Performance Center, Washington D.C., District of Columbia
  - Orthopedic Center of Palm Beach City, Atlantis, Florida
  - Baptist Health Orthopedic Care - Miami Gardens, Maimi, Florida
  - Infinite Clinical Research, Miami, Florida
  - Gulfcoast Research Institute, Sarasota, Florida
  - Clinical Research of West Florida, Tampa, Florida
  - Hospital for Special Services, West Palm Beach, Florida
  - Injury Care Research, Boise, Idaho
  - Kansas City Bone & Joint Clinic - Overland Park, Overland Park, Kansas
  - Ochsner Sports Medicine Institute, New Orleans, Louisiana
  - New England Baptist Hospital, Boston, Massachusetts
  - Oakland Medical Center, Troy, Michigan
  - Sundance Clinical Research, St Louis, Missouri
  - New York-Presbyterian Queens, Flushing, New York
  - West Clinical Research, Morehead City, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Ohio State University, Columbus, Ohio
  - University Orthopedics Center, Altoona, Pennsylvania
  - Altoona Arthritis & Osteoporosis Center - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - University Orthopedics Center (UOC) - State College, State College, Pennsylvania
  - Medical University Health - West Ashley Medical Pavilion, Charleston, South Carolina
  - Texas Orthopedic Specialists, PLLC, Bedford, Texas
  - First Surgical Hospital, Bellaire, Texas
  - El Paso Clinical Trials, LLC, El Paso, Texas
  - Physicians Research Options, Draper, Utah
  - Spectrum Medical, Danville, Virginia